CLINICAL TRIAL: NCT01437189
Title: Clinical Protocol of Self-Controlled Study on the Effects of Sertraline on Depression in Parkinson's Disease
Brief Title: The Effects of Sertraline on Depression in Parkinson's Disease
Acronym: PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Wei Luo, associate professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WS1851055
Record Dates: First submitted 2011-09-16; First posted 2011-09-20 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Depression; Parkinson's Disease
Keywords: Parkinson's disease; depression; sertraline; intervention
MeSH Terms: conditions — Depression; Parkinson Disease | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Parkinson's disease patients with depression (Experimental): It is a self-controlled study only contains one arm, aims to investigate the effects of Sertraline on depression in Parkinson's disease
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — Starting dose 25mg/day for 1 week, then increasing to 50mg/day, add on 50mg each time when the depressive symptoms are not improved, at 2-week intervals. Maximum: 200mg/day. Maintenance: lowest effective dose.
  Other Names: Zoloft

SUMMARY:
The aim of this open-label, self-control study is to evaluate the efficacy of sertraline in treating depression in Patients with Parkinson's disease. In addition, the investigators also want to find out whether patient gets better quality of life when depression is improved.

DETAILED DESCRIPTION:
Depression in PD is associated with more severe cognitive and functional impairments, a faster progression of illness, worse quality of life, increase mortality and higher burden for caregivers, when compare PD patients without depression. Depression accounts for approximately 40-50% in PD patients, which is also well known as a main factor impacting on health-related quality of life (HRQoL) in negative way in the context of PD and even their caregivers. In our previous cross-sectional study, the investigators have already studied the prevalence of depressive symptoms in PD patients and also have proved how depressive symptoms severely worsen HRQoL in PD patients in the area of the mainland China. In order to improve HRQoL of PD, some interventions, for example, taking some antidepressants to improve depression are urgently required. In addition, the investigators had already tested the validity and reliability of Chinese version of the 39-item Parkinson's disease questionnaire (PDQ-39) in mainland China, the paper about which already have been published in journal of Zhejiang university science B (biomedicine and biotechnology) already, therefore, the investigators can use the questionnaire of Chinese version of PDQ-39 to assess PD patients' quality of life.

Treatment of depression with antidepressant drugs is well established. In the last 20 years, the application of antidepressant has risen mainly due to the introduction of the selective serotonin reuptake inhibitors (SSRIs). These drugs are now the most commonly prescribed antidepressants in patients with depression in general. Regarding depression in the context of PD, a recent survey in the U.S. showed that 63% of the prescriptions for depression in PD were for SSRIs and only 7.5% for tricyclic antidepressants (TCAs). The preference of SSRIs over the older TCAs is supposedly based on their similar efficacy but better tolerability, especially when compared with tertiary amines, such as amitriptyline or imipramine. Sertraline is characterized by a low selectivity for serotonin relative to dopamine reuptake, suggesting a favorable efficacy profile. There was a randomized study pointing out that both sertraline and low-dose amitriptyline improved depressive symptoms in PD, and a significant benefit on quality of life was observed only with sertraline. Still, more studies are needed to demonstrate whether sertraline is effective to depression in PD patients. Further more, there is no trial about the efficacy and safety of sertraline on depression in PD in mainland China. It's necessary for us to initiate and conduct this trial in mainland China.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 35 and 75 years of age from the outpatients clinic in Department of Neurology, the Second Affiliated Hospital, School of Medicine, Zhejiang University.
2. All patients should have a confirmed diagnosis of PD according to Brain Bank Criteria.
3. Diagnosed to be major depression episode according to DSM-IV,
4. Mini Mental State Examination (MMSE) exclude dementia.

Exclusion Criteria:

1. Mini-Mental State Examination (MMSE) demonstrate dementia
2. Any current DSM-IV Axis I diagnosis other than a depressive or anxiety disorder.
3. History of psychosis or hallucinations or under treatment with atypical neuroleptics.
4. Treatment-resistant depression. Treatment-resistant depression (TRD) occurs when a patient with unipolar depression fails to respond to adequate antidepressant therapy.
5. Pregnancy or lactation.
6. Concomitant use in patients taking monoamine oxidase inhibitors (MAOIs).
7. Concomitant use in patients taking pimozide.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2013-08-01 (Actual); Study Completion 2013-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Luo, PH.D&M.D, Principal Investigator — School of medcine, Zhejiang University
Locations (1):
- Department of Neurology, the Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Marino S, Sessa E, Di Lorenzo G, Digangi G, Alagna A, Bramanti P, Di Bella P. Sertraline in the treatment of depressive disorders in patients with Parkinson's disease. Neurol Sci. 2008 Dec;29(6):391-5. doi: 10.1007/s10072-008-1021-3. Epub 2008 Nov 11. PMID 19002650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start on August/01 2011 Location: the second affiliated hospital of Zhejiang University, School of medicine.
Groups:
- Parkinson's Disease Patients With Depression: This arm received treatment of Sertraline. Sertraline: Starting dose 25mg/day for 1 week, then increasing to 50mg/day, add on 50mg each time when the depressive symptoms are not improved, at 2-week intervals. Maximum: 200mg/day. Maintenance: lowest effective dose.
Period: Overall Study
Arm/Group | Parkinson's Disease Patients With Depression
Started | 35
Completed | 20
Not Completed | 15
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 4
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | Parkinson's Disease Patients With Depression
Number analyzed (Participants) | 35
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 60 [43 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 20
Region of Enrollment [Count of Participants; unit: Participants]
  China | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Depression Rating Scale (HAMD)
Description: The minimum and maximum value of HAMD is 0 and 96 respectively. The higher score means worse severity of depression.
  Combined with reducing scores rate of HAMD, there are four grades: heal (HAMD is lower than 8 or reducing rate is higher than 75%), excellent utility (reducing rate is between 50% and 75%), utility (reducing rate is between 25% and 50%) and nullity (reducing rate is lower than 25%).
Time Frame: baseline, 8 weeks (endpoint)
Measure: Median (Standard Error); unit: score on a scale
Groups:
- Parkinson's Disease Patients With Depression: This arm received treatment of Sertraline. Sertraline: Starting dose 25mg/day for 1 week, then increasing to 50mg/day, add on 50mg each time when the depressive symptoms are not improved, at 2-week intervals. Maximum: 200mg/day. Maintenance: lowest effective dose.
  after 8 weeks. the score of Hamilton Depression Rating Scale was compared.
Arm/Group | Parkinson's Disease Patients With Depression
Number analyzed (Participants) | 20
score on a scale
  baseline | 48.1 (7.4)
  endpoint | 35.5 (10.5)

2. Secondary Outcome: Change From Baseline in Questionnaire of PDQ-39,
Description: The minimum and maximum value of PDQ-39 is 0 and 116respectively. The higher score means worse severity of quality of life.
Time Frame: Baseline, 8 weeks (endpoint)
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Parkinson's Disease Patients With Depression
Number analyzed (Participants) | 20
units on a scale
  baseline | 51 (10.5)
  endpoint | 46 (9.7)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each visit from administration to endpoint.
Arm/Group | Parkinson's Disease Patients With Depression
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 3/35
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parkinson's Disease Patients With Depression (N=35)
dizziness (Nervous system disorders) | 2 (2) — one patient took 50mg and another one took 75mg and developed dizziness.
nausea (Gastrointestinal disorders) | 1 (1) — the patient developed nausea when he took 75mg sertraline

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No